CLINICAL TRIAL: NCT05470127
Title: Evaluation of the Performance of a Novel Prostate Biopsy System Compared With Standard of Care Biopsy Needle on Quantitative and Qualitative Tissue Parameters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uro-1 Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SUREcore v. SOC
Record Dates: First submitted 2022-07-11; First posted 2022-07-22 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Prostate Disease; Prostate CA
Keywords: Prostate CA; Needle biopsy
MeSH Terms: conditions — Prostatic Diseases

STUDY DESIGN:
Intervention Model Description: The two biopsy needle sets will be used in the same patient during the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SUREcore biopsy needle (Experimental): The SUREcore needle will be used to collect up to 10 tissue samples
  Interventions: Device: Prostate biopsy needle
- Standard of Care biopsy needle (Active Comparator): The urologist will use his/her standard biopsy needle to collect up to 15 tissue samples
  Interventions: Device: Prostate biopsy needle

INTERVENTIONS:
Device: Prostate biopsy needle — Prostate tissue biopsy with a biopsy needle

SUMMARY:
Currently used biopsy devices do not predictably obtain full cores of tissue and the tissue obtained is often fragmented and disrupted making it difficult for pathological review. This post-market study will assess the utility of the SUREcore biopsy needle and the coreCARE specimen retrieval device versus a standard of care biopsy needle and the typical tissue container used in urology offices and clinics today.

DETAILED DESCRIPTION:
The safety and performance of the SUREcore and coreCARE devices will be compared to matched prostate tissue collected with a standard of care biopsy needle and tissue retrieval system. Following informed consent, prostate tissue biopsy samples will be obtained using the systematic 12 core biopsy template-- 6 with the typical biopsy needle and 6 with the SUREcore needle. Tissue samples will be randomized to retrieval with the swiping method or using the coreCARE device. Adverse events will be documented both during the procedure and within 5 days after the procedure. The user will be asked to rank the use of both biopsy tools during the procedure and a pathologist will be asked to assess the quality of the tissue cores obtained.

ELIGIBILITY:
Inclusion Criteria:

* Adult male scheduled for prostate biopsy
* Able to provide informed consent
* Able and willing to provide verbal assessment of his condition 5 days post-procedure

Exclusion Criteria:

* Unwilling to provide consent

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate tissue is to be collected, which is only present in males.
Enrollment: 200 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Procedure Success | 1 Day of the procedure
  Percentage of tissue samples collected that are suitable for pathological review
Core length of tissue in the sample | 1 Day of the procedure
  Quantity of Tissue Samples Collected
weight of tissue in the sample | 1 Day of the procedure
  Quantity of Tissue Samples Collected
Tissue Sample Preparation | 1 Day of the procedure
  Time required to prepare the tissue samples for pathological review

SECONDARY OUTCOMES:
Ease of use of the biopsy needle | 1 Day of the procedure
  Utility of the biopsy needle measured with a Likert scale of 1 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lawson, PhD, Study Director — Lawson & Associates
Locations (1):
- Georgia Urology, Cartersville, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Likert scale means for use of either of the biopsy needles will be available upon request